CLINICAL TRIAL: NCT03798899
Title: Multicentre, Randomised, Double-blind Study Assessing the Efficacy and Safety of Penthrox® Combined With a Standard Analgesia (SoC) in Comparison to a Placebo Combined With a Standard Analgesia (SoC) in Adult Patients Admitted to the Emergency Department With Moderate to Severe Pain Associated With Trauma
Brief Title: Efficacy and Safety of Penthrox® Combined With a Standard Analgesia (SoC) in Adult Patients Admitted to the Emergency Department With Moderate to Severe Pain Associated With Trauma
Acronym: Pen ASAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma SAS (Industry)
Collaborators: AXONAL (Unknown); Exystat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MR311-4501; 2017-004469-28 (EudraCT Number)
Record Dates: First submitted 2018-11-09; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Methoxyflurane; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Penthrox® (Methoxyflurane) (Experimental): Patients will be asked to inhale Penthrox® intermittently or continuously to obtain adequate analgesia.
  Penthrox® or placebo will be administered in combination with standard analgesic treatments usually used according to the emergency department protocol (SoC).
  Duration of treatment: 1 administration (with a maximum of 2 inhalers) during passage to emergency.
  Interventions: Drug: Methoxyflurane
- Normal Saline (Placebo Comparator): Patients will be asked to inhale Penthrox® intermittently or continuously to obtain adequate analgesia.
  Penthrox® or placebo will be administered in combination with standard analgesic treatments usually used according to the emergency department protocol (SoC).
  Duration of treatment: 1 administration (with a maximum of 2 inhalers) during passage to emergency.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Methoxyflurane — PENTHROX 3mL inhalation vapour, liquid
  Other Names: Penthrox®
  Arms: Penthrox® (Methoxyflurane)
Drug: Normal Saline — Placebo
  Arms: Normal Saline

SUMMARY:
A phase 4 randomised, double-blind study to assess the efficacy and safety of Penthrox® used from the outset in multimodal analgesia, in combination with the standard analgesic protocol used in the department, for conscious adult patients presenting in an emergency department with moderate to severe pain associated with a trauma

DETAILED DESCRIPTION:
On admission, the patient pain score will be measured using a numerical scale (NRS-11) to verify the eligibility of the patient in the study (NRS ≥ 4).

At the time of randomisation, the patient's pain score will be measured using a VAS in order to verify the patient's eligibility for randomisation (VAS ≥ 40).

Admissible patients will be randomised by IWRS (Interactive Web Response System) to receive:

* Either Penthrox® + SoC
* Or placebo + SoC (Figure 1). Randomisation will be stratified by sex, site and according to the baseline pain score (NRS 4-5 for a moderate-intensity pain versus NS 6-10 for a severe-intensity pain).

The IWRS system will be based on the fact of including 50% patients with moderate pain and 50% patients with severe pain.

Close weekly monitoring of this ratio will be set up. The decision to no longer include patients in one of the study subgroups according to pain, if necessary, or to change this ratio, will be made by the Study Sponsor and in agreement with the study investigator-coordinator and the study scientific committee. A minimum of 150 patients will be included in the severe pain subgroup (EN 6-10).

The treatment (preparation of two inhalers, the second only being given to the patient on request) will only be administered once intermittently or continuously to patients on admission to the study (D0, T0).

The pain score will be assessed using the VAS every 5 minutes up to 20 minutes, then at 30, 60, 90, and 120 minutes after the start of study treatment (T0). Patients will be assessed until their discharge from the emergency departments (hospitalization, transfer home, transfer to the operating room) or up to 120 minutes after the initial administration.

A telephone interview will take place 14 (± 2) days after the first treatment administration to assess the medium-term safety of the product.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older
* Patients (in an emergency, parent or relative) who dated and signed their informed consent to participate in the study
* Patients admitted to the emergency department due to a trauma
* Patients having a pain score ≥ 4 measured using a numerical scale (NRS) at the time of admission to emergency departments.
* Patients having a pain score ≥ 40 measured using the VAS at the time of randomisation.

Exclusion Criteria:

* Life-threatening conditions requiring immediate admission to the operating theatre or the intensive care unit;
* Impaired consciousness according to the investigator regardless of the cause, including head trauma or drug or alcohol consumption;
* Acute medicinal or alcohol intoxication, according to the investigator;
* Pregnant woman or woman at risk of pregnancy and not using highly effective contraception methods or known lactation;
* Analgesic treatment within 5 hours (8 h for sodium diclofenac) prior to admission, except for paracetamol, which is allowed;
* Treatment with nitrous oxide within 5 hours before presentation at the emergency department;
* Use of analgesics for chronic pain;
* Prior use of Penthrox®;
* Use of an investigational product one month before presentation at the emergency department;
* Hypersensitivity to Penthrox® or any other fluoridated anesthetic;
* History of signs of hepatic lesions after use of methoxyflurane or after anaesthesia by a halogenated hydrocarbon;
* Malignant hyperthermia: Known malignant hyperthermia or patient genetic predisposition or patient or family history of serious adverse reactions;
* Clinical evidence of respiratory depression according to the investigator;
* Clinical evidence of cardiovascular instability according to the investigator;
* Clinical renal or hepatic damage, according to the investigator, pre-existing or known;
* Presence of any other clinical condition that can, according to the investigator's opinion, have an impact on the patient's ability to participate in the study or the results of the study.
* Individuals protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
time until pain relief defined by the duration between the start of the study treatment (T0) and pain relief | through study completion, maximum of 2 hours
  Measured on Pain intensity visual analogue scale (PI-VAS) 0-100 where 100 is the highest pain

SECONDARY OUTCOMES:
Duration between the start of study treatment (T0) and pain relief reported by the patient | through study completion, maximum of 2 hours
  Pain measured on PI-VAS, 0-100 where 100 is the highest pain
Absolute Pain Intensity Difference (PID) measured using the PI-VAS at 5, 10, 15, 20 and 30 minutes after T0 | baseline to 5, 10, 15, 20 and 30 minutes
  PID for a given assessment time is equal to the VAS score at T0 minus the VAS score at each assessment time provided in the study. Pain measured on PI-VAS, 0-100 where 100 is the highest pain
Relative Pain Intensity Difference measured using the PI-VAS at 5, 10, 15, 20 and 30 minutes after T0 | baseline to 5, 10, 15, 20 and 30 minutes
  Relative pain intensity difference for a given assessment time is equal to the VAS score at T0 minus the VAS score at each assessment time provided in the study divided by the VAS score at T0. Pain measured on PI-VAS, 0-100 where 100 is the highest pain
Pain relief defined by pain intensity < 40 mm on the PI-VAS scale at 5, 10, 15, 20 and 30 minutes after T0 | baseline to 5, 10, 15, 20 and 30 minutes
  Pain measured on PI-VAS, 0-100 where 100 is the highest pain
Response defined by pain reduction of 20 mm on the PI-VAS at 5, 10, 15, 20 and 30 minutes after T0 | baseline to 5, 10, 15, 20 and 30 minutes
  Pain measured on PI-VAS, 0-100 where 100 is the highest pain
Response defined by pain reduction of 30% mm on the PI-VAS at 5, 10, 15, 20 and 30 minutes after T0 | baseline to 5, 10, 15, 20 and 30 minutes
  Pain measured on PI-VAS, 0-100 where 100 is the highest pain
Summed Pain Intensity Difference (SPID) measured on the PI-VAS at 5, 10, 15, 20 and 30 minutes | baseline to 30 minutes
  SPID will be calculated by using the pain intensity difference (PID) at each of these assessment times provided in the study. SPID is the sum of the PID at each study assessment time, weighted by using the time elapsed since the previous assessment, and approaches the area under the curve for the PID over time. Relative to the VAS score, the SPID measurement has the advantage of considering individual differences at the level of initial pain intensity (baseline) as well as time.
Proportion of patients attaining an SPID of at least 33% | through study completion, maximum of 2 hours
  The proportion of patients attaining an SPID of at least 33% of the maximum possible SPID will be calculated (maximum possible SPID is the the value that would be obtained if the patient was pain free (VAS=0) for the entire study period); this will be considered as corresponding to the responder rate. A % SPID of 33% was previously established as being a clinically significant measurement in pain results.
Quantity of opioids received (in milligrams of morphine) | through study completion, maximum of 2 hours
Description of the Standard of Care and concomitant analgesic treatments | through study completion, maximum of 2 hours
  Descriptions from the World Health Organization (http://www.who.int/cancer/palliative/painladder/en/): Type of drug, doses, administration periods, and treatment duration
Sedation score (Ramsay scale) | through study completion, maximum of 2 hours
  Measured using the Ramsay sedation scale
Patient satisfaction score (Likert 0-5 scale) | through study completion, maximum of 2 hours
  Satisfaction is rated by patient as Poor, Fair, Good, Very Good or Excellent
Physician satisfaction scale (Likert 0-5 scale) | through study completion, maximum of 2 hours
  Satisfaction is rated by Physician as Poor, Fair, Good, Very Good or Excellent
Nurse satisfaction scale (Likert 0-5 scale) | through study completion, maximum of 2 hours
  Satisfaction is rated by Nurse as Poor, Fair, Good, Very Good or Excellent
Length of stay (LOS) in emergency | through study completion, maximum of 2 hours
Assess the time until medical decision to discharge | through study completion, maximum of 2 hours
Incidence of adverse events (AE) not associated with the underlying trauma and occurring during treatment | through study completion, maximum of 2 hours
Change in blood pressure | baseline to 30 minutes
  The Blood Systolic and Diastolic pressure (mmHg) will be measured at baseline and 30 minutes. The difference between the values will be calculated.
Change in oxygen saturation | baseline to 30 minutes
  Oxygen saturation (%) will be measured at baseline and 30 minutes. The difference between the values will be calculated.
Change in respiration rate | baseline to 30 minutes
  Respiration rate (breaths/min) will be measured at baseline and 30 minutes. The difference between the values will be calculated.
Change in heart rate | baseline to 30 minutes
  Heart rate (beats/min) will be measured at baseline and 30 minutes. The difference between the values will be calculated.
Incidence of tachycardia, hypotension, hypertension and respiratory depression | through study completion, maximum of 2 hours
Incidence of premature withdrawal of patients for safety or tolerability reasons | through study completion, maximum of 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: A Ricard-Hibon, Dr, Principal Investigator — CHG Pontoise / SAMU 95
Locations (8):
- France (8):
  - CH Annecy Genevois, Annecy
  - GH Carnelle Porte de l'Oise, Beaumont-sur-Oise
  - Hôpital Avicenne - APHP, Bobigny
  - CHRU Lille, Lille
  - Hôpital Edouard Herriot, Lyon
  - Hospice civil de Lyon, Pierre-Bénite
  - CH René Dubos, Pontoise
  - CHU Purpan, Toulouse